CLINICAL TRIAL: NCT06088745
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial to Evaluate the Protective Efficacy, Safety, and Immunogenicity of Recombinant Herpes Zoster Vaccine (CHO Cells) in Subjects Aged 40 Years and Older
Brief Title: A Phase Ⅲ Clinical Study to Evaluate Protective Efficacy and Safety of a Recombinant Herpes Zoster Vaccine
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Luzhu Biotechnology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LZ901-300
Record Dates: First submitted 2023-09-26; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Vaccine-Preventable Diseases; Herpes Zoster
MeSH Terms: conditions — Vaccine-Preventable Diseases; Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment main group (Experimental): 11500 subjects in treatment main group will receive 2 doses of LZ901 at D0 and D29. This group will be required to complete a 12 month safety follow-up after full immunization.
  Interventions: Biological: Recombinant Herpes Zoster Vaccine
- Placebo main group (Placebo Comparator): 11500 subjects in placebo main group will receive 2 doses of placebo at D0 and D29. This group will be required to complete a 12 month safety follow-up after full immunization.
  Interventions: Biological: Recombinant Herpes Zoster Vaccine Placebo
- Treatment immunization group (Experimental): 1500 subjects in treatment immunization group will receive 2 doses of LZ901 at D0 and D29. This group is designed to evaluate the batch-batch immunogenicity consistency among three different batches of LZ901, as well as the immunogenicity and immunogenicity persistence of the LZ901 at 36 months after full immunization.
  Interventions: Biological: Recombinant Herpes Zoster Vaccine
- Placebo immunization group (Placebo Comparator): 1500 subjects in placebo immunization group will receive 2 doses of placebo at D0 and D29. This group is designed to evaluate the batch-batch immunogenicity consistency among three different batches of LZ901, as well as the immunogenicity and immunogenicity persistence of the LZ901 at 36 months after full immunization.
  Interventions: Biological: Recombinant Herpes Zoster Vaccine Placebo

INTERVENTIONS:
Biological: Recombinant Herpes Zoster Vaccine — The active ingredient of the recombinant herpes zoster vaccine is varicella-zoster virus glycoprotein E fusion protein expressed in CHO cells by gene recombination technology. The LZ901 cell line carrying this gene is cultured in chemically defined medium. The harvest cell culture is purified by multi-step liquid chromatography. After Low pH incubation and virus removal filter package Nanofiltration inactivation/virus removal process, the bulk containing high-purity recombinant herpes zoster virus glycoprotein E is obtained. Finally, an alumina adjuvant is added to the formulated final product.
  Other Names: LZ901
  Arms: Treatment immunization group; Treatment main group
Biological: Recombinant Herpes Zoster Vaccine Placebo — Alumina adjuvant
  Arms: Placebo immunization group; Placebo main group

SUMMARY:
This clinical trial is to study protective efficacy and safety of a recombinant herpes zoster vaccine (LZ901) and sponsored by Beijing Luzhu Biotechnology Co., Ltd. It is a phase Ⅲ, randomized, double-blind, placebo-controlled in healthy people aged 40 years and older. The study is to protect adults against shingles (herpes zoster / varicella zoster virus(VZV)). There will be about 26000 participators who will receive two-dose injection at the upper arm.

LZ901 vaccine is made up of a tetramer of VZV glycoprotein E (VZV gE-Fc) and adsorbed with aluminum hydroxide adjuvant. This adjuvant can raise the immune response to a lot of antigens. It is the most widely used and safe adjuvant in various types of vaccines worldwide.

DETAILED DESCRIPTION:
In this study:

1. The participation is voluntary.
2. Before the trial, participants will receive some tests for screening. If qualified, investigators will officially invite them to join this trial.
3. The trial vaccine is LZ901 (100μg/0.5 mL). The placebo, which is aluminum hydroxide adjuvant, has no active drug. Participants will receive one of two as above mentioned.
4. This trial included a protective efficacy test and a batch-to-batch consistency test (immunization subgroup). Approximately 26000 subjects aged 40 years and older will be enrolled. Subjects will be randomized to receive either LZ901 or placebo in which about 3000 subjects will be enrolled into immunization subgroup and randomly receive three different batches LZ901 and one batch placebo at a ratio of 1:1:1:3. The immunization subgroup was designed to evaluate the batch-batch immunogenicity consistency among three different batches of LZ901, as well as the immunogenicity and immunogenicity persistence of the LZ901 at 12, 24, and 36 months after full immunization.
5. All subjects will receive the LZ901 or Placebo on day 0 and day 29. Subject will have 16 visits, including 5 on-site visits and 11 in-person visits except for subjects in the immunization subgroup who have 24 visits, including 8 on-site visits and 16 in-line visits.
6. The primary objective was to evaluate the Vaccine Efficacy (VE) of LZ901 against herpes zoster, as compared with placebo, after 30 days of full immunization in people 40 years of age and older.
7. The secondary objective was to evaluate the protective efficacy of LZ901, as compared with placebo, against laboratory-confirmed cases of HZ after 30 days of full vaccination in people 40 years of age and older. To evaluate the safety of LZ901. The immunogenicity of LZ901was evaluated (immunization subgroup). To evaluate the batch-to-batch consistency of immunogenicity of three batches of LZ901 in subject aged ≥40 years (immunization subgroup).
8. An exploratory objective was to evaluate the effect of LZ901 on reducing the severity of PHN in HZ subjects ≥40 years old." To evaluate the efficacy of LZ901 compared with placebo in preventing PHN in subjects ≥40 years old with HZ efficacy endpoint. The immunogenicity of LZ901 was evaluated at 12, 24 and 36 months after full immunization in subject ≥40 years old (immunization subgroup).

ELIGIBILITY:
Inclusion Criteria:

* Males and females able to provide legal identity certificate, aged ≥ 40 years inclusive at the time of signing the ICF;
* Able to understand the study procedures, voluntarily agree to participate in the study, and sign the ICF;
* Female subjects are not pregnant or lactating. Female subjects with childbearing potential should take reliable contraceptive measures, and have no pregnancy and fertility plan within 7 months;
* Axillary temperature ≤ 37.0℃ on the day of enrollment;
* Able to attend all scheduled follow-up visits and able to comply with protocol requirements;

Exclusion Criteria:

* Subjects who have had herpes zoster within the previous 5 years;
* Previous vaccination against varicella or shingles (including use of a registered product or participation in a clinical trial of varicella or shingles vaccine);
* Hypersensitivity to any of the components of the test vaccine: or prior hypersensitivity to any recombinant vaccine of CHO cell origin [e.g., recombinant hepatitis B vaccine (CHO cell)], polysorbate, etc.; or prior history of severe allergy* to any of the vaccinations;

  *Severe allergies: anaphylaxis, anaphylactic laryngeal edema, anaphylactic purpura, thrombocytopenic purpura, localized anaphylactic necrotic reaction (Arthus reaction), severe urticaria.
* Developed immunodeficiency diseases (congenital or acquired immunodeficiency diseases, human immunodeficiency virus infection) or received immunosuppressive/cytotoxic treatments (cancer chemotherapy, organ transplantation, or treatment planned during a clinical trial in the 6 months prior to vaccination);
* Receiving immunosuppressive therapy (e.g., long-term systemic glucocorticoid application for ≥14 days at a dose of ≥2 mg/kg/day or ≥20 mg/day of prednisone or prednisone-equivalent dose) within 3 months prior to vaccination or within 1 month after the planned full course of immunization；
* Received an inactivated or recombinant vaccine or mRNA vaccine within 14 days or any live attenuated vaccine within 28 days prior to vaccination;
* Subjects who are suffering from an acute illness or are in the acute exacerbation phase of a chronic disease within 3 days prior to vaccination;
* History of asplenia or functional asplenia, and asplenia or splenectomy due to any condition;
* Treatment with blood products or globulins within 3 months prior to enrollment, or planned use of such products within 2 months of vaccination;
* Participating in other clinical studies of investigational or un-registered products (drugs, vaccines or devices, etc.), or planning to participate in other clinical studies before the end of this clinical study;
* Significant underlying medical conditions that, in the opinion of the investigator, may prevent completion of the trial (e.g., life-threatening disease that may limit survival to less than 4 years) or any other condition

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The Vaccine Efficacy | 30 days after full immunization
  To evaluate the Vaccine Efficacy in the prevention of HZ compared to placebo based on the number of confirmed cases of HZ

SECONDARY OUTCOMES:
Solicited AE | from 0 to 7 days after each dose
  Incidence of Solicited AE include site of vaccination (local) and non-site of vaccination (systemic)
Unsolicited AE | From 0 to 30 days after each dose
  Incidence of unsolicited AEs, include all AEs, except solicited AEs reported Days 0~6 after the study intervention.
AE | Within 30 minutes after each dose
  Incidence of AE refers to any untoward medical occurrence in a subject administered the investigational vaccine.
Adverse Events of Special Interest | From initial dose to 30 days after full immunization
  Confirmed cases of HZ within 30 days after the first dose and full immunization
Serious Adverse Event | From first dose to 12 months after full immunization
  The incidence of all serious adverse events (SAEs)
Anti-GE antibody | 30 days after full immunization
  Seroconversion rate of anti-GE antibody in three different batches of immunization groups
Geometric Mean Fold Increase | 30 days after full immunization
  Geometric Mean Fold Increase (GMFI) of anti-GE antibody in three different batches of immunization groups compared with pre-vaccination (day 0)
GMC ratios | 30 days after full immunization
  GMC ratios of anti-GE antibodies in three different batches of immunization groups

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, MM, Principal Investigator — Jiangsu Province Center for Disease Control and Prevention (China)
Locations (1):
- Jiangsu Province Center for Disease Control and Prevention (China), Zhenjiang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No